CLINICAL TRIAL: NCT00539526
Title: Evaluation of Hyperemia With the Use of Ocular Prostaglandin Analogues
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-LUM-07-003
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): bimatoprost 0.03%
  Interventions: Drug: Bimatoprost 0.03%
- 2 (Active Comparator): travoprost 0.004%
  Interventions: Drug: travoprost 0.004%
- 3 (Active Comparator): latanoprost 0.005%
  Interventions: Drug: latanoprost 0.005% eye drops

INTERVENTIONS:
Drug: Bimatoprost 0.03% — bimatoprost 0.03%, 1 drop nightly for 3 months
  Other Names: Lumigan®
  Arms: 1
Drug: travoprost 0.004% — travoprost 0.004% eye drops, 1 drop nightly for 3 months
  Other Names: Travatan® Z
  Arms: 2
Drug: latanoprost 0.005% eye drops — latanoprost 0.005%, 1 drop nightly for 3 months
  Other Names: Xalatan®
  Arms: 3

SUMMARY:
This study will evaluate hyperemia and ocular surface tolerability in patients on prostaglandin analogues

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma (pseudoexfoliative or pigmentary glaucomas are allowed) or ocular hypertension

Exclusion Criteria:

* Known contraindication to latanoprost, bimatoprost or travoprost
* Uncontrolled systemic disease
* Active ocular disease other than glaucoma or ocular hypertension
* Pregnant or lactating women or women of childbearing potential NOT utilizing a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Diego, California, United States

REFERENCES:
- [Background] Whitson JT, Trattler WB, Matossian C, Williams J, Hollander DA. Ocular surface tolerability of prostaglandin analogs in patients with glaucoma or ocular hypertension. J Ocul Pharmacol Ther. 2010 Jun;26(3):287-92. doi: 10.1089/jop.2009.0134. PMID 20578283

RESULTS

PARTICIPANT FLOW:
Groups:
- Bimatoprost 0.03%: bimatoprost 0.03%
- Travoprost 0.004%: travoprost 0.004%
- Latanoprost 0.005%: latanoprost 0.005%
Period: Overall Study
Arm/Group | Bimatoprost 0.03% | Travoprost 0.004% | Latanoprost 0.005%
Started | 35 | 33 | 38
Completed | 32 | 31 | 36
Not Completed | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.03% | Travoprost 0.004% | Latanoprost 0.005% | Total
Number analyzed (Participants) | 35 | 33 | 38 | 106
Age, Continuous [Mean (Full Range); unit: years] | 69.3 [57 to 81] | 65.4 [52 to 78] | 67.3 [57 to 77] | 67.3 [52 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 19 | 61
  Male | 13 | 13 | 19 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Conjunctival Hyperemia Scores at Month 3
Description: Change from baseline in mean conjunctival hyperemia scores at month 3. Hyperemia is engorgement of the blood vessels (redness) of the bulbar conjunctiva of the eye (the clear membrane covering the white surface of the eye). Hyperemia was graded using a 5-point scale in which 0=no redness and +3=deep, diffuse redness. A negative number change from baseline indicates improvement.
Time Frame: Baseline, Month 3
Measure: Mean (Standard Error); unit: Scores on Scale
Arm/Group | Bimatoprost 0.03% | Travoprost 0.004% | Latanoprost 0.005%
Number analyzed (Participants) | 35 | 33 | 38
Scores on Scale
  Baseline | 0.74 (0.10) | 0.86 (0.12) | 0.74 (0.11)
  Month 3 | 0.05 (0.1) | 0.07 (0.13) | 0.06 (0.10)

2. Secondary Outcome: Change From Baseline in Corneal Staining With Fluorescein at Month 3
Description: Change from baseline in corneal staining with fluorescein at month 3. The cornea is the transparent front part of the eye which covers the iris and pupil. To detect the presence or absence of corneal puncta (tiny disruptions in the surface of the eye), fluorescein dye is administered into the eye and the eye is graded using a 5-point scale where 0 equals no puncta (best), and 3 equals too many puncta to count (worst). A negative number change from baseline indicates improvement.
Time Frame: Baseline, Month 3
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Bimatoprost 0.03% | Travoprost 0.004% | Latanoprost 0.005%
Number analyzed (Participants) | 35 | 33 | 38
Scores on a Scale
  Baseline | 0.59 (0.12) | 0.48 (0.11) | 0.70 (0.13)
  Month 3 | 0.15 (0.15) | -0.07 (0.12) | -0.18 (0.11)

3. Secondary Outcome: Change From Baseline in Tear Break-Up Time (TBUT) at Month 3
Description: Change from baseline in TBUT at month 3. TBUT is defined as the time (seconds) required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. A positive number change from baseline indicates improvement.
Time Frame: Baseline, Month 3
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Bimatoprost 0.03% | Travoprost 0.004% | Latanoprost 0.005%
Number analyzed (Participants) | 35 | 33 | 38
Seconds
  Baseline | 9.1 (1.0) | 7.9 (0.8) | 8.6 (0.8)
  Month 3 | 0.5 (0.9) | 1.7 (0.8) | 0.4 (1.0)

ADVERSE EVENTS:
Arm/Group | Bimatoprost 0.03% | Travoprost 0.004% | Latanoprost 0.005%
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33 | 0/38
Other Adverse Events (participants affected / at risk) | 1/35 | 2/33 | 0/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03% (N=35) | Travoprost 0.004% (N=33) | Latanoprost 0.005% (N=38)
Headache (Nervous system disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo